CLINICAL TRIAL: NCT06860997
Title: Clinical Echocardiography and S' Wave for Early Recognition of Acute Coronary Syndrome in the Emergency Department, A Prospective Study
Acronym: CLEAR_ECHO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024/28OCT/476
Record Dates: First submitted 2025-02-28; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction (MI); Non-ST Elevation Myocardial Infarction; Unstable Angina; Echocardiography; Tissue Doppler; Emergency Medicine; Cardiac Function Tests
Keywords: Acute Coronary Syndrome (ACS); Non-ST Elevation Myocardial Infarction (NSTEMI); Unstable Angina; Tissue Doppler Imaging (TDI); Echocardiography; S' wave velocity; Mitral Annular Plane Systolic Excursion (MAPSE); Tricuspid Annular Plane Systolic Excursion (TAPSE); Emergency Medicine; Diastolic function; Point-of-Care Ultrasound (PoCUS); Bedside Echocardiography; Cardiac Function Assessment; Early ACS Detection; Regional Wall Motion Abnormalities; Diagnostic Accuracy
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Echocardiographic Assessment for Early ACS Detection (Other): This arm involves bedside echocardiographic assessment using tissue Doppler imaging (TDI) S' wave velocity to evaluate its diagnostic accuracy for acute coronary syndrome (ACS) in patients presenting with acute chest pain in the emergency department (ED).
  Interventions: Diagnostic Test: Tissue Doppler Imaging (TDI) S' Wave Echocardiography

INTERVENTIONS:
Diagnostic Test: Tissue Doppler Imaging (TDI) S' Wave Echocardiography — This intervention involves bedside echocardiographic assessment using TDI S' wave velocity to evaluate its diagnostic accuracy for acute coronary syndrome (ACS) in patients presenting with acute chest pain in the emergency department (ED).

SUMMARY:
The goal of this prospective observational study is to assess the diagnostic accuracy of the tissue Doppler imaging (TDI) S' wave in detecting acute coronary syndrome (ACS) in adult patients presenting to the emergency department (ED) with acute chest pain. This study focuses on patients aged 18 years or older, who require continuous cardiac monitoring but do not show ST-elevation myocardial infarction (STEMI) on their initial ECG.

The main questions it aims to answer are:

* Can TDI S' wave velocity serve as an early diagnostic marker for ACS in the emergency department?
* How does the diagnostic performance of TDI S' compare with other echocardiographic markers (MAPSE, TAPSE, and diastolic parameters such as E, E', A, E/A, E/E')?
* Do demographic factors (age, sex, BMI, echogenicity) influence the diagnostic accuracy of echocardiographic parameters for ACS? If there is a comparison group: Researchers will compare TDI S' wave velocity findings with the final adjudicated diagnosis of ACS (determined after 3 months) to evaluate its sensitivity and specificity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Presenting to the emergency department (ED) with acute chest pain
* No ST-elevation myocardial infarction (STEMI) on initial ECG
* Requiring continuous cardiac monitoring based on triage decision
* Able to provide informed consent (written consent required)

Exclusion Criteria:

* Known pre-existing cardiomyopathy (e.g., hypertrophic cardiomyopathy, dilated cardiomyopathy)
* Severe valvular heart disease
* Left bundle branch block (LBBB) or presence of a pacemaker
* Arrhythmias (e.g., atrial fibrillation, frequent premature ventricular contractions)
* Cardiac arrest or cardiogenic shock at presentation
* Pulmonary hypertension
* Pericardial effusion or tamponade
* Non-cardiac cause of chest pain suspected as the primary diagnosis
* Language barrier preventing informed consent (study materials available in English, French, and Dutch)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of Tissue Doppler Imaging (TDI) S' Wave for Acute Coronary Syndrome (ACS) Diagnosis | 3 months
  The study will assess the diagnostic accuracy (sensitivity and specificity) of TDI S' wave velocity in detecting ACS in patients presenting to the emergency department (ED) with acute chest pain.
  The reference standard for comparison will be the final ACS diagnosis, determined by an adjudication committee based on a review of medical records, ECG findings, cardiac biomarkers (troponins), and follow-up assessments at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Bastian Rodrigues de Castro, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium